CLINICAL TRIAL: NCT01276678
Title: Multi-Analyte, Genetic, and Thrombogenic Markers of Atherosclerosis (The MAGMA STUDY)
Brief Title: Multi-Analyte, Genetic, and Thrombogenic Markers of Atherosclerosis
Acronym: MAGMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: Accumetrics, Inc. (Industry); Nanosphere, Inc. (Industry)
Responsible Party: Principal Investigator, Kevin Bliden, Sinai Center for Thrombosis Research Program Manager, LifeBridge Health
Other Study IDs: 1478
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biomarker Analysis by Multi-Analyte Profiling Genetic Testing-GWAS and CYP2C19 genotyping Comprehensive Lipoprotein Cholesterol Profile Platelet aggregation and Thrombelastography-Clot characteristics and antiplatelet response Urinary 11-dehydrothromboxane
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: 300 healthy controls free from any pharmacologic therapy
- Suspected CAD - Cardiac Cathetrization: subject's ≥18 years undergoing coronary angiography (inpatient cohort)or who have undergone coronary angiography within 5 years

SUMMARY:
About 13 million people in the United States have coronary artery disease (CAD). It is the leading cause of death in both men and women.

Coronary artery disease (CAD) occurs when the blood vessels that supply blood to the heart muscle (the coronary arteries) become hardened and narrowed. The arteries harden and narrow due to buildup of fatty and calcified material called plaque on their inner walls. The buildup of plaque is also called atherosclerosis. This is a process which starts early in life, but can be influenced by multiple factors.

Several factors increase the risk of developing atherosclerosis. They include high blood pressure, smoking, diabetes, high cholesterol and being related to someone who had a heart attack or a stroke. The more risk factors you have, the greater the chance that you have severe atherosclerosis. Some of the risk factors cannot be modified, like age and family history of early heart disease. The influenceable factors include high blood pressure, high blood cholesterol, high blood sugar, cigarette smoking, overweight or obesity, and lack of physical activity.

Nevertheless, there are patients without any above mentioned risk factors who develop atherosclerosis. In addition to that, there are also patients with several risk factors who do not develop severe coronary artery disease.

According to research studies high blood levels of some substances in the blood (biochemical markers) as well as some genes in the DNA of our cells may be associated with an increased risk of developing CAD and faster progression of the disease.

The purpose of this study is to find a correlation between certain blood markers and growth of the plaques, regardless of the presence of the classic risk factors for atherosclerosis. If we prove our hypothesis we will be one step closer to predicting the extent of atherosclerosis by performing certain blood tests.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD), primarily coronary artery disease are the leading cause of death and disability in the United States and Europe. The cost of cardiovascular disease in the United States in 2009 is estimated to be $475.3 billion, according to the American Heart Association and the National Heart, Lung, and Blood Institute. Although there have been significant accomplishments in reducing cardiovascular events over the past decade, too many people still die of heart and vascular diseases. Therefore, the improvement of risk stratification of CVD by identification of new biomarkers has been extensively investigated in both primary and secondary clinical settings in the past decade. A substantial number of biomarkers, representing various stages of atherogenesis and impaired cardiac function, have been evaluated against modifiable traditional risk factors, such as cholesterol, blood pressure, smoking status, and diabetes. However, little is known about the true extent that these identified multi-analyte, genetic, and thrombogenic markers contribute to the presence and degree of atherosclerosis.

Patients with severe stenosis of coronary arteries may have a different profile of biochemical and genetic markers than patients with "clear" coronary vessels. Therefore, more research is required to improve the predictability and specificity of these known and novel factors before physicians fully implement these tests into their routine clinical practice.

At present, physicians rely on conventional cardiovascular risk factors to try to identify at-risk patients. A number of risk factors stem from genetic or biologic conditions such as gender, age, ethnicity and family history of heart disease. While many risk factors cannot be changed, risk factors such as high cholesterol, high blood pressure, obesity, tobacco smoking, stress, physical inactivity can be modified. One of the most significant risk factor for the development of CVD is diabetes mellitus, whereby both heredity and lifestyle play a major role. Nevertheless, there are patients without these known classical risk factors who develop severe CVD. Conversely, there are patients with these classical risk factors without relevant coronary artery disease. "The CVD Risk Factor Paradox" may be explained by a combination of biological, environmental, and genetic factors that are under investigation.

Animal and human studies have established the role of cholesterol in the development and progression of atherosclerosis. Epidemiological studies directly implicated LDL-C to the development of atherosclerosis and CVD. Furthermore, LDL-C level appears to be directly related to the development and recurrence of CVD. While LDL-C is the primary lipid marker for assessing risk, evidence has demonstrated the important role of other lipoproteins components in atherogenesis. These include lipoprotein (a), LDL pattern density, HDL subtypes, VLDL, and intermediate-density lipoprotein. A substantial body of evidence has also demonstrated Lp-PLA2 as a cardiovascular risk marker in both primary and secondary prevention that provides new information, over and above new traditional risk factors. Most recently oxidized low-density lipoprotein (oxLDL)/ β2-glycoprotein I (β2GPI) complexes have been implicated in atherogenesis. More accurate and expanded depiction of the lipid profile compared to the standard lipid profile may identify important emerging risk factors and secondary targets of therapy for cardiovascular disease.

It is also been established that heightened plaque metabolism together with increased blood vulnerability characterized by hypercoagulability, heightened platelet reactivity and inflammation, are important processes responsible for plaque rupture and subsequent occlusive ischemic events occurrence during ACS. Recent developments in catheter-based near-infrared spectroscopy may help to identify vulnerable plaques by characterizing chemical components. However, information regarding blood vulnerability based on a specific biomarker profile is lacking.

Multiple lines of evidence suggest the critical role of platelets in the development of atherosclerosis and thrombosis. By expressing adhesion molecules platelets facilitate the diapedesis of leukocytes into the vascular wall during atherosclerotic development. Additionally, P-selectin and CD40L trigger release of RANTES from platelets and subsequently augment monocyte recruitment and secretion of inflammatory cytokines from monocytes. Previous studies have demonstrated the roles of MCP-1 and IL-8 during plaque development and cardiovascular clinical outcomes. Gurbel et. al. demonstrated that incremental changes in platelet function, demonstrated by increases in GPIIb/IIIa expression and increased release of RANTES, IL-8 and MCP-1, as clinical disease progressed from the asymptomatic state to stable angina and finally to unstable angina.These findings further reinforce the critical role of platelets in plaque destabilization.

The role of inflammation during atherosclerotic plaque rupture and subsequent development of thrombus generation at the site of plaque rupture by enhancing tissue factor expression and thrombin generation is well recognized. Several studies have demonstrated the association of high IL-6, -8, and -18, elevated CD40 ligand (CD40L), myeloperoxidase, tumor necrosis factor and CRP levels with ischemic events.

Epidemiological evidence in addition to experimental and clinical data supports the hypothesis that CRP may be a "marker" as well as an active participant in the development of atherothrombotic complications. More interestingly, recent in vitro studies suggest that there is a direct role of CRP on endothelial and platelet function. In autopsy studies, CRP immune reactivity was detected in atherosclerotic arteries but not in normal arteries. In addition, the levels of CRP in fibrous tissue and atheroma of atherectomy specimens were higher in patients with unstable angina and myocardial infarction compared to patients with stable angina. Gurbel et al. demonstrated a statistically significant increase in specific inflammation markers, importantly CRP, IL-8, RANTES and MCP-1 in patients with progressive CAD compared to patients with asymptomatic disease. Although serial changes in markers were not studied in the same patient, the incremental changes among various markers across the study population, clearly suggests the transition between disease states.

Linking vulnerable blood characterized by elevated inflammation markers, hypercoagulability, and highly reactive platelets to the vulnerable patient who is at risk for thrombotic complications has been the subject of much discussion in recent years.

Platelet activation and aggregation are the most critical factors in the generation of ischemic events, including stent thrombosis and myocardial infarction (MI). Unlike the routine measurement of blood glucose, cholesterol and C-reactive protein performed during the management of patients with atherosclerosis, the measurement of platelet function is largely ignored during the management of cardiovascular patients, even in those at the highest risk. Multiple laboratory and translational research studies performed at our research center as well as others have demonstrated the importance of platelet reactivity as a new emerging risk factor. At our center we primarily utilize two methods to determine coagulation and platelet reactivity, thrombelastography (TEG) and platelet aggregation. The indications for TEG testing include assessing bleeding of unclear etiology, and assessing hypercoagulable states. In addition, TEG platelet mapping has been utilized to monitor antiplatelet therapy. It has been hypothesized that high platelet-fibrin clot strength measured by TEG predicts robust clot formation at the site of plaque rupture. In support of this premise, Gurbel et al. demonstrated that high thrombin-induced platelet-fibrin clot strength and high platelet reactivity has been associated with ischemic events in patients with CVD. In fact, all of the current data support that uniform measurement of on-treatment platelet reactivity may be a major diagnostic strategy, not only in the treatment of patients who have undergone PCI, but also in all patients with cardiovascular disease at risk for thrombotic events.

Presently, the gold standard to diagnose patients with CVD is coronary angiography. If significant lesions are detected, coronary intervention with angioplasty or coronary artery bypass grafting can be performed to reestablish flow in the blocked coronary arteries. Modification of cardiovascular risk factors and pharmacological management is subsequently implemented to prevent recurrent cardiovascular events including myocardial infarction and stent thrombosis. The importance of the ADP-P2Y12 receptor interaction and COX-inhibition has been demonstrated by the clinical benefits associated with the addition of clopidogrel to aspirin therapy in patients with acute coronary syndromes and patients treated with stents. However, the" one size fits all" antiplatelet management strategy has proven to be flawed due to clopidogrel and aspirin response variability.

Incomplete inhibition of platelet thromboxane generation has been associated with an increased risk of cardiovascular events. In the CHARISMA study, Eikelboom et. al. demonstrated that urinary concentrations of 11-dehydro thromboxane B2 potentially was a modifiable determinant of stroke, myocardial infarction, or cardiovascular death in patients at risk for atherothrombotic events. In addition, variability in clopidogrel response is well established with multiple translational research studies demonstrating a relationship between antiplatelet nonresponsiveness, high on-treatment platelet reactivity, and the occurrence of ischemic events in percutaneous coronary intervention patients.

Recently, the loss-of-function CYP2C19*2 allele has been shown to be associated with decreased activation of clopidogrel and antiplatelet effect and with increased cardiovascular events in patients receiving clopidogrel. Individuals with this genotype have reduced protection from thrombotic events as outlined in the FDA black box warning for clopidogrel. Despite the black box warning, there has been no large scale study performed to personalize antiplatelet treatment of P2Y12 inhibitors with CYP2C19 genotyping primarily because the technology for point-of-care genotyping is not commercially available. From a clinical perspective, reporting 2C19 test results in a rapid fashion will help guide therapeutic decisions while patients are in the inpatient setting prior to discharge.

Large-scale genome-wide association studies using high-density, single nucleotide polymorphism genotyping arrays have revealed genetic variants that are robustly associated with CAD and CAD-related traits such as type 2 diabetes and obesity. Also, evidence has been obtained that multiple rare alleles with fairly strong phenotypic effects may contribute to the genetic heritability of CAD Although, the involvement of specific genes and their level of contribution to CAD have not been established by research, it is known that CAD often results from the blended effects of multiple genes. These so-called polygenic effects mean that the genetics of CAD are extremely complicated, with many different genes influencing person's risk. In most cases, CAD is not inherited in a clearly dominant or recessive manner. Instead, a person may have mutations in some genes that increase risk and mutations in other genes that decrease risk, and their combined effect plays a role in the development of atherosclerosis. At present the replication of results in the reported studies is poor, probably because of the lack of high-quality environmental data and not counting for the gene-environment interactions.

Many patients have undetected coronary artery disease that, if accurately identified, would lead to more aggressive early treatment strategies, including lifestyle modification and targeted pharmacologic therapy. A goal of current study is to determine potential biochemical and genetic markers associated with the presence and progression of CVD.

The current studies hypothesis is that specific biomarkers and genetic profile will precisely identify with the severity of angiographically-defined coronary lesions, independently of the classic risk factors for atherosclerosis. The investigators believe that this will enhance the treatment of patients with cardiovascular disease by implementing personalized treatment strategies.

3. STUDY DESIGN 3.1. Outline A total of 1300 subject's ≥18 years undergoing coronary angiography (inpatient cohort)or who have undergone coronary angiography within 5 years (outpatient cohort, not to exceed 50 subjects) will be enrolled. In addition, 300 healthy controls free from any pharmacologic therapy will also be enrolled. After giving informed consent, a lifestyle questionnaire on topics of diet, physical activity, history of high blood pressure, hyperlipidemia, diabetes, smoking and family history of early heart disease will be completed. A blood (approximately 35 ml) and urine sample will be obtained prior to angiogram for the inpatient cohort, or on the day of enrollment for the outpatient cohort for laboratory assessments. The presence and severity of CAD will be determined according to the following three categories: category 1 - no disease or minimal stenosis (<25%) of major branches without need of any medical therapy; category 2 - intermediate stenosis (25%-75%) of major branches and/or patient needs only conservative treatment (no need for PTCA); category 3 - severe stenosis (>75%) of major branch and/or patient needs PTCA or CABG. Statistical tools will be used to detect any correlation between the studied markers and the extent of atherosclerotic plaques. Subgroup analysis will be performed to detect the similar correlation in certain risk groups like smokers, obese subjects, diabetes, or subjects with hypercholesterolemia. Subjects will be contacted once a year for up to 5 years by telephone and information regarding antiplatelet therapy and cardiovascular events (death, myocardial infarction, stent thrombosis, stroke, revascularization, major bleeding) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Subjects scheduled for coronary angiography
* Subjects who have undergone coronary angiography within 5 years

Exclusion Criteria:

* Female subjects who are pregnant
* Subjects who suffer currently from an acute infection
* Subjects, who have received an experimental drug or who gave a blood donation of ≥ 1 pint within 8 weeks prior to screening
* Subjects with any coagulation, bleeding or blood disorders
* Subjects who are undergoing treatment for neoplastic diseases
* Subjects with autoimmune disease or connective tissue disease
* Subjects with HIV or hepatitis C.
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with the interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 1300 subject's ≥18 years undergoing coronary angiography (inpatient cohort)or who have undergone coronary angiography within 5 years (outpatient cohort, not to exceed 50 subjects) will be enrolled. In addition, 300 healthy controls free from any pharmacologic therapy will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
severity of angiographically-defined coronary lesions as determined by comprehensive biomarker risk profile | 1.5 years
  To develop a comprehensive biomarker risk profile that will correlate with the severity of angiographically-defined coronary lesions, independently of the classic risk factors for atherosclerosis.

SECONDARY OUTCOMES:
Genetic Components | 5 years
  To evaluate the contribution of genetic components to the presence of coronary artery disease in association with environmental factors. Of interest is to see whether certain genes might accelerate atherosclerosis in subgroups like smokers, diabetics, obese subjects, or various ethnic groups
Biomarker Profile | 1.5 years
  To determine the difference in the biomarker profile between CAD patients, patients with no known angiographically identified disease and healthy volunteers.
Drug treatment strategies | 1.5 years
  To determine the effect of different drug treatment strategies on biomarker profile.
Prediction Model | 1.5 years
  To create prediction model for major CV events based on genetic and other nongenetic biomarkers.
Verigene | 1.5 years
  To demonstrate the utility of the Point-of-Care Verigene 2C19/CBS Nucleic Acid Assay for detecting CYP2C19 variants.
Urinary 11-dehydro thromboxane B2 | 1.5 years
  To determine an association between urinary 11-dehydro thromboxane B2 concentrations with the severity of angiographically-defined coronary lesions.
Lp-PLA2 | 1.5 years
  To determine the association between Lp-PLA2 and angiographically-defined coronary lesions.
Association of low-density lipoproteins/β2-glycoprotein I (β2GPI) | 1.5 years
  To determine the association between oxidized low-density lipoprotein (oxLDL)/ β2-glycoprotein I (β2GPI) complexes and angiographically-defined coronary lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, M.D., FACC, Principal Investigator — Sinai Center for Thrombosis Research
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bliden KP, Singla A, Gesheff MG, Toth PP, Tabrizchi A, Ens G, Guyer K, Singh M, Franzese CJ, Stapleton D, Tantry US, Gurbel PA. Statin therapy and thromboxane generation in patients with coronary artery disease treated with high-dose aspirin. Thromb Haemost. 2014 Aug;112(2):323-31. doi: 10.1160/TH14-01-0094. Epub 2014 Apr 24. PMID 24763965